CLINICAL TRIAL: NCT05328076
Title: Analysis of Parathyroid Vascularization During Total Thyroidectomy Using Quantitative Real-time Indocyanine Green Angiography
Brief Title: Parathyroid Vascularization During Total Thyroidectomy Using Indocyanine Green Angiography
Acronym: ANGIO_PARA
Status: Terminated | Type: Observational
Why Stopped: We encountered problems in finding the necessary resources in the Institute
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Riccardo Maggiore, Principal Investigator, IRCCS San Raffaele
Other Study IDs: ANGIO PARA
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Thyroid; Thyroid Cancer; Hypoparathyroidism; Vascularization
Keywords: Parathyroid; Thyroid surgery; Indocyanine green angiography
MeSH Terms: conditions — Thyroid Diseases; Thyroid Neoplasms; Hypoparathyroidism; Neovascularization, Pathologic | interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Surgical group: Patients who undergo thyroid surgery and receive indocyanine green angiography
  Interventions: Drug: Indocyanine green; Device: SPY Portable Handheld Imaging (SPY-PHI)

INTERVENTIONS:
Drug: Indocyanine green — Indocyanine green is used to perform intraoperative angiography.
Device: SPY Portable Handheld Imaging (SPY-PHI) — The device is used to perform intraoperative angiography.

SUMMARY:
Prospective, observational, single-center study about the use of indocyanine green angiography during total thyroidectomy.

The main objective of the study is to identify a quantitative score of parathyroid vascularization as an outcome of angiography that correlates with the absence of postoperative hypoparathyroidism.

It is planned to enroll 66 patients.

DETAILED DESCRIPTION:
Postoperative hypoparathyroidism and subsequent hypocalcemia are the most frequent complications after thyroid surgery. The incidence ranges from 19-38%, depending on the definition of hypoparathyroidism and hypocalcemia.

Although the cause of postoperative hypoparathyroidism is multifactorial, one of the most important factors is vascularization of parathyroid glands left in situ that is insufficient or impaired by surgical manipulation. Therefore, one of the goals of thyroid surgery is not only to recognize the parathyroid glands during dissection but also to respect their vascularization in order to preserve well perfused and viable glands.

The general objective of this study is to quantitatively assess the vascularization of the parathyroids following total thyroid removal.

In particular, the investigators intend to obtain data regarding parathyroid vascularization during total thyroidectomy with indocyanine green angiography. During standard surgery, angiography will be performed using a special camera after having administered intravenously indocyanine green. This technique is used to objectively assess the degree of fluorescence of the parathyroid glands.

ELIGIBILITY:
Inclusion Criteria:

* Able to sign informed consent
* Indication to total thyroidectomy
* No contraindication to indocyanine green administration

Exclusion Criteria:

* Evidence of parathyroid disease
* Allergy to iodinated contrast
* Chronic kidney failure
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients who need surgical treatment for thyroid disease.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Vascularization score | Intraoperatively
  A quantitative score of parathyroid vascularization as an outcome of indocyanine green angiography during thyroidectomy that correlates with the absence of postoperative hypoparathyroidism.
  The score will be reported as a percentage (range 0% - 200%) where the higher score means the better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Rosati, Prof., Study Director — San Raffaele Hospiral
Locations (1):
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lang BH, Wong CK, Hung HT, Wong KP, Mak KL, Au KB. Indocyanine green fluorescence angiography for quantitative evaluation of in situ parathyroid gland perfusion and function after total thyroidectomy. Surgery. 2017 Jan;161(1):87-95. doi: 10.1016/j.surg.2016.03.037. Epub 2016 Nov 10. PMID 27839936
- [Background] Vidal Fortuny J, Sadowski SM, Belfontali V, Guigard S, Poncet A, Ris F, Karenovics W, Triponez F. Randomized clinical trial of intraoperative parathyroid gland angiography with indocyanine green fluorescence predicting parathyroid function after thyroid surgery. Br J Surg. 2018 Mar;105(4):350-357. doi: 10.1002/bjs.10783. Epub 2018 Feb 6. PMID 29405252
- [Background] Spartalis E, Ntokos G, Georgiou K, Zografos G, Tsourouflis G, Dimitroulis D, Nikiteas NI. Intraoperative Indocyanine Green (ICG) Angiography for the Identification of the Parathyroid Glands: Current Evidence and Future Perspectives. In Vivo. 2020 Jan-Feb;34(1):23-32. doi: 10.21873/invivo.11741. PMID 31882459
- [Background] Puzziello A, Rosato L, Innaro N, Orlando G, Avenia N, Perigli G, Calo PG, De Palma M. Hypocalcemia following thyroid surgery: incidence and risk factors. A longitudinal multicenter study comprising 2,631 patients. Endocrine. 2014 Nov;47(2):537-42. doi: 10.1007/s12020-014-0209-y. Epub 2014 Feb 22. PMID 24563161
- [Background] Ji YB, Song CM, Sung ES, Jeong JH, Lee CB, Tae K. Postoperative Hypoparathyroidism and the Viability of the Parathyroid Glands During Thyroidectomy. Clin Exp Otorhinolaryngol. 2017 Sep;10(3):265-271. doi: 10.21053/ceo.2016.00724. Epub 2016 Aug 13. PMID 27515510
- [Background] Zaidi N, Bucak E, Yazici P, Soundararajan S, Okoh A, Yigitbas H, Dural C, Berber E. The feasibility of indocyanine green fluorescence imaging for identifying and assessing the perfusion of parathyroid glands during total thyroidectomy. J Surg Oncol. 2016 Jun;113(7):775-8. doi: 10.1002/jso.24237. Epub 2016 Apr 4. PMID 27041628